CLINICAL TRIAL: NCT00308789
Title: Infant Flow Biphasic NCPAP Versus Infant Flow NCPAP for the Facilitation of Successful Extubation in Infants </= 1250 Grams: A Randomized Controlled Trial
Brief Title: A Trial of Infant Flow Biphasic Nasal Continuous Airway Pressure (NCPAP) Versus Infant Flow NCPAP for the Facilitation of Extubation in Infants </= 1250 Grams
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-0258-A
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Infant, Premature, Diseases; Bronchopulmonary Dysplasia; Apnea of Prematurity
Keywords: Continuous Positive Airway Pressure; Infant,newborn; Artificial respiration
MeSH Terms: conditions — Infant, Premature, Diseases; Bronchopulmonary Dysplasia; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Biphasic NCPAP
  Interventions: Procedure: Biphasic Infant flow NCPAP
- 2 (Active Comparator): Continuous CPAP
  Interventions: Procedure: CPAP

INTERVENTIONS:
Procedure: Biphasic Infant flow NCPAP — Biphasic Nasal continuous positive airway pressure
  Arms: 1
Procedure: CPAP — Continuous positive airway pressure
  Arms: 2

SUMMARY:
The purpose of this study is to compare two methods of delivering Nasal Continuous Airway Pressure (NCPAP): Biphasic Mode and a continuous mode, to see which is better in getting babies off the ventilator and decreasing lung damage.

DETAILED DESCRIPTION:
Chronic lung disease (CLD) remains a significant problem among low birth weight infants with a reported incidence of up to 26% in infants < 1500 grams. Nasal continuous positive airway pressure (NCPAP) has been demonstrated to provide effective non-invasive respiratory support for preterm infants. The use of NCPAP is associated with a decreased need for mechanical ventilation and may impact on the incidence of CLD. There are two types of NCPAP now available, a Biphasic mode which allows for cycling at two different levels of positive pressure and a continuous mode which allows only for one level of positive pressure.

Comparisons: Biphasic NCPAP will be compared with continuous CPAP to see which better facilitates the extubation of preterm infants who weigh </= 1250 grams at birth. The incidence of CLD, retinopathy of prematurity, sepsis, intraventricular haemorrhage, periventricular leucomalacia and necrotizing entercolitis will also be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Infants </= 1250 grams who are going to be extubated

Exclusion Criteria:

* Congenital abnormalities of the upper airway
* Acquired nasal septum injury
* Congenital Heart Disease excluding Patent Ductus arteriosus

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The rate of successful extubation with either mode of NCPAP | Day 7 post primary extubation

SECONDARY OUTCOMES:
The incidence of chronic lung disease
The incidence of other complications of prematurity including sepsis,retinopathy of prematurity, intraventricular haemorrhage/periventricular leucomalacia and necrotizing entercolitis
The predictive value of the minute ventilation test

CONTACTS AND LOCATIONS:
Overall Officials: Karel O'Brien, MB, FRCPC, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] O'Brien K, Campbell C, Brown L, Wenger L, Shah V. Infant flow biphasic nasal continuous positive airway pressure (BP- NCPAP) vs. infant flow NCPAP for the facilitation of extubation in infants' </= 1,250 grams: a randomized controlled trial. BMC Pediatr. 2012 Apr 4;12:43. doi: 10.1186/1471-2431-12-43. PMID 22475409